CLINICAL TRIAL: NCT00196612
Title: Phase II Randomized Trial Comparing Efficacy and Safety of the Maintenance of a HAART Association Protease Inhibitor Containing Versus a Once Daily Antiretroviral Triple Association, in HIV Adult Patients With Undetectable Viral Load.ANRS 099 ALIZE
Brief Title: Once Daily Antiretroviral Therapy in HIV Infected Adults Treated With HAART
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Triangle Pharmaceuticals (Industry); Gilead Sciences (Industry); Bristol-Myers Squibb (Industry); Dupont Applied Biosciences (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 099 ALIZE
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: HIV Infections
Keywords: HIV Infections; Reverse Transcriptase Inhibitors; Treatment simplification
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine; Racivir; Pharmaceutical Preparations; Didanosine; efavirenz

INTERVENTIONS:
Drug: emtricitabine, FTC (drug)
Drug: didanosine, ddI (drug)
Drug: efavirenz (drug)

SUMMARY:
The combination of two nucleoside analogues and one protease inhibitor is a highly active antiretroviral therapy (HAART) in HIV infected adults. In those with an undetectable viral load, a once daily combination of FTC, ddI, efavirenz would be easier to take, with less side effects and the same efficacy. The aim of the study was to evaluate if the once daily combination presents the same efficacy than the HAART therapy with less side effects and a better adherence.

DETAILED DESCRIPTION:
The combination of two nucleoside analogues and one protease inhibitor is a highly active antiretroviral therapy (HAART) in HIV infected adults, but side effects an the great number of pills induces less adherence to the therapy. Once daily combination with a lower number of pills could be more easy to take, with a greater adherence, less side effects, and the same efficacy. 355 patients are recruited in the study, randomized in two treatment groups: maintenance of the HAART therapy versus changing for a once daily combination of FTC, ddI, efavirenz, during 48 weeks. The primary end-point is the viral success maintained until 48 weeks. Secondary end-point is the safety and adherence.

The trial is prolonged for a total of 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected adults
* Antiretroviral treatment since 6 months, with two nucleoside analogues and one or two protease inhibitors
* CD4 cell count over 100/mm3
* HIV RNA below 400 copies/ml since 6 months
* Signed written informed consent

Exclusion Criteria:

* Previous treatment with non nucleoside analogue, ddI alone
* Pregnancy
* Alcool abuse
* Acute infection, past neurological or pancreatic disease, biological abnormalities
* Chemotherapy or immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 2001-04; Study Completion 2004-09

PRIMARY OUTCOMES:
Virological success from W0 to W48

SECONDARY OUTCOMES:
Progression of HIV infection
CD4 cell count
Safety
Treatment adherence
Quality of life
Viral mutations
Therapeutic strategy failure

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Molina, MD, PhD, Principal Investigator — Service de Maladies Infectieuses, Hôpital Saint-Louis, Paris, 75475, France; Genevieve Chene, MD, PhD, Study Director — INSERM unité 593, Bordeaux, France

REFERENCES:
- [Result] Molina JM, Journot V, Morand-Joubert L, Yeni P, Rozenbaum W, Rancinan C, Fournier S, Morlat P, Palmer P, Dupont B, Goujard C, Dellamonica P, Collin F, Poizot-Martin I, Chene G; ALIZE (Agence Nationale de Recherches sur le SIDA 099) Study Team. Simplification therapy with once-daily emtricitabine, didanosine, and efavirenz in HIV-1-infected adults with viral suppression receiving a protease inhibitor-based regimen: a randomized trial. J Infect Dis. 2005 Mar 15;191(6):830-9. doi: 10.1086/428091. Epub 2005 Feb 10. PMID 15717256